CLINICAL TRIAL: NCT07301619
Title: Post-marketing Clinical Investigation to Evaluate the Efficacy and Safety of BtHCROSS for Restoring Facial Volume and Filling Facial Folds and Wrinkles
Brief Title: Post-market Study on BtHCROSS® for Restoring Facial Volume After a Single Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i+Med S.Coop. (Industry)
Collaborators: Dr. Goya Análisis, SL. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BtHCROSS-PIC01-2021
Record Dates: First submitted 2025-11-27; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Aesthetics Procedure
Keywords: hyaluronic acid; crosslinking; skin rejuvenation; facial volume restoration; facial wrinkle and folds; soft tissue augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BtHCROSS® (Experimental): Single injection of 1 ml of viscoelastic sodium hyaluronate solution crosslinked
  Interventions: Device: BtHCROSS®

INTERVENTIONS:
Device: BtHCROSS® — Single injection of 1 ml of viscoelastic sodium hyaluronate solution crosslinked

SUMMARY:
This clinical study investigated the safety and effectiveness of BtHCROSS, a hyaluronic acid-based injectable used to restore facial volume and reduce wrinkles. Adults aged 30 to 70 received a single treatment and were monitored over 9 months. Researchers assessed improvements in facial appearance and recorded any side effects. The results aimed to support the product's continued safe use in aesthetic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 30 and 70 years.
* Individuals showing mild to moderate signs of facial skin aging (such as loss of brightness, hydration, and/or firmness).
* Sufficient willingness and ability, as judged by the investigator, to complete the study questionnaires.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Known allergy or sensitivity to hyaluronic acid or any other ingredient in the product.
* Individuals who have undergone any wrinkle correction or rejuvenation procedures in the past 6 months or during the study (e.g., radiofrequency, electrotherapy, botulinum toxin, thread lifts, or laser techniques).
* Autoimmune or inflammatory diseases, or any condition affecting skin health that could interfere with the treatment.
* History of any illness or infection in the injection area during the study.
* Lymphatic and/or vascular disorders.
* Individuals with unrealistic expectations about the treatment outcomes.
* Previous facial surgery.
* Active infection in the treatment area.
* Blood coagulation disorders. Subjects on anticoagulant therapy are excluded, even without a diagnosed coagulation issue, unless cleared by their prescribing specialist.
* Subjects with unrealistic expectations regarding the likely outcomes of the treatment.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Determine the BtHCROSS' efficacy in improving the facial volume loss | 6 months
  To determine how effective BtHCROSS is in improving volume loss in the mid-face region comparing the skin's condition before and after treatment. This evaluation is carried out by medical professionals using validated aesthetic scales, depending on the specific product model. The measurements were done using the MFVLS (Mid-Face Volume Loss Scale) a 0-5 scale, 0 being good outcome and 5 being the worst outcome.
Determine the BtHCROSS' efficacy in improving facial wrinkle severity | 6 months
  To determine how effective BtHCROSS is in improving wrinkle severity comparing the skin's condition before and after treatment. This evaluation is carried out by medical professionals using validated aesthetic scales, depending on the specific product model. The measurements were done using the WSRS(Wrinkle Severity Rating Scale) a 0-5 scale, 0 being good outcome and 5 being the worst outcome.
Determine the BtHCROSS' efficacy in improving lip fullness | 6 months
  To determine how effective BtHCROSS is in improving vlip fullness comparing the lips's condition before and after treatment. This evaluation is carried out by medical professionals using validated aesthetic scales, depending on the specific product model. The measurements were done using the LFGS (Lip Fullness Grading Scale) a 0-5 scale, 0 being good outcome and 5 being the worst outcome.
Safety Outcome | 9 months
  The study evaluates the safety of BtHCROSS by systematically recording and analyzing any serious adverse events that occur during the treatment period.

SECONDARY OUTCOMES:
Exploratory objective - Global Aesthetic Improvement Scale (GAIS) by investigator | 6-9 months
  To assess overall aesthetic improvement using the Global Aesthetic Improvement Scale (GAIS), a widely used 5-point Likert scale ranging from "Exceptional Improvement" (5) to "Worsening" (1). This measurements were done by the investigator.
Exploratory objective - Subjective self assessment of the treatment by the patient | 6-9 months
  After the final treatment session, each participant self-assessed their perceived improvement through a likert-type 5 point brief questionnaire, which answers were (worsening, no changes, improvement, important improvement and exceptional improvement)

CONTACTS AND LOCATIONS:
Locations (1):
- Complutense Medical Center (Virtus Group), Madrid, Madrid, Spain